CLINICAL TRIAL: NCT06944873
Title: Metabolic Reprogramming of Monocytes in Inflammatory Flares of Inflammatory Bowel Diseases
Acronym: REPRO-MICI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institute for Advanced Biosciences (IAB), Grenoble (Unknown)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0363
Record Dates: First submitted 2025-01-13; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Monocytes; Metabolic reprogramming
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood test 4 EDTA tubes — Blood test 4 EDTA tubes for biological check-up

SUMMARY:
Inflammatory bowel diseases, Crohn's disease and haemorrhagic rectocolitis, are pathologies that progress in flare-ups, impacting on patients' quality of life and functional or even vital prognosis. These inflammatory diseases require the use of immunosuppressive and immunomodulatory treatments, the side-effects of which can be significant, and the limited number of which sometimes puts patients and practitioners in a therapeutic impasse from which surgery is the only way out. It is therefore important to be able to develop new therapeutic approaches, ideally better tolerated, that can control inflammation during relapses. Monocytes are one of the main players in the inflammatory reaction. In the laboratory, we have developed a strategy for the metabolic reprogramming of these cells based on the use of oxygen microbubbles to modulate the inflammatory response of monocytes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18
* Managed at the CHUGA for a severe IBD flare-up requiring hospitalisation or endoscopy for flare-up
* Patient not objecting to the REPRO-MICI study

Exclusion Criteria:

* Patients protected by law (pregnant or breast-feeding women, minors, patients under guardianship or trusteeship, persons deprived of their liberty or hospitalised under duress).
* Patients with positive HIV, HBV or HCV serology.
* Patients with a positive ELISPOT with no history of treatment for latent tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IBD in severe relapse requiring hospitalisation for immunosuppressive therapy or endoscopy for relapse.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-16 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparaison of reduction of concentration of inflammatory cytokines and chemokines in cells treated by oxygen microbubbles vs cells not treated | up to 2 years
  Validation of inhibition of the production of inflammatory cytokines and chemokines by the monocytes treated by oxygen microbubbles

SECONDARY OUTCOMES:
Comparaison of tissue factor expression at the membrane of monocytes treated by microbubbles vs monocytes not treated | up to 2 years
  Inhibition of tissue factor expression at the membrane of treated monocytes
Comparaison of glucose metabolism rate in monocytes treated bu microbubbles vs not treated cells | up to 2 years
  Modulation of glucose metabolism in treated monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Marianne HUPE, MD PhD, Principal Investigator — Grenoble Alpes University Hospital
Locations (1):
- Grenoble Alpes University Hospital, La Tronche, France

IPD SHARING:
Plan to Share IPD: No